CLINICAL TRIAL: NCT04098315
Title: Registro Italiano Dei Pazienti Con Infezione da HIV-1 Con RESistenza Agli Inibitori Della Trascrittasi Inversa, Dell'InteGrasI e Della PrOteasi Virale (PRESTIGIO)
Brief Title: Italian Registry of HIV-1 Infected Patients With Drug-RESistant Virus to Reverse Transcriptase Inhibitors, InteGrasE and Viral Protease.
Acronym: PRESTIGIO
Status: Recruiting | Type: Observational
Sponsor: Castagna Antonella (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Castagna Antonella, Sponsor and Principal Investigator, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: PRESTIGIO
Record Dates: First submitted 2019-09-16; First posted 2019-09-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: HIV-1-infection; Multi-Antiviral Resistance
Keywords: HIV; AIDS; DRUG RESISTANCE
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — At enrolment, plasma and cell samples of peripheral blood mononuclear cells(PBMCs) are collected for subsequent virological and immunological investigations. The samples to be collected for each patient are: 6 plasma aliquots (1.5-2.0 ml/each) and 6 PBMC aliquots (3-5 million/each).
  Sample collection should be repeated at the end of each subsequent year of follow-up.
  The collected biological samples are sent to the biobank of the coordinating centre and stored in a biological bank with ISO 9001:2000 quality certification (Biorep srl, http://www.biorep.it/).
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: REGISTER CREATION — Build a national registry of patients with HIV-1 infection and documented resistance to the 4 classes of antiretroviral drugs.

SUMMARY:
The PRESTIGIO Registry is an Observational, prospective, multicentre study that includes patients, regularly followed by Italian Infectious Disease Centres, with HIV-1 infection and documented resistance to the 4 classes of antiretroviral drugs: nucleoside reverse transcriptase inhibitors (NRTI), non-nucleoside reverse transcriptase inhibitors (NNRTI), protease inhibitors (PI), and integrase inhibitors (INSTI).

Main objective of this register is to evaluate in the study population:

* the long-term effectiveness of different antiretroviral regimes;
* evolution of the genotype and phenotypic susceptibility of antiretroviral drugs used in patients with virological failure;
* mortality;
* incidence of opportunistic AIDS-related infections and chronic conditions (comorbidity);
* determinants of clinical outcomes including virological/immunological/inflammatory markers.
* antiretroviral therapy (ART) compliance and health assessments;
* drug-economy indications related to the clinical management of this complex sub-population.

DETAILED DESCRIPTION:
The PRESTIGIO Register consists of a systematic and continuous collection of data on clinical, laboratory and treatment characteristics of patients with documented resistance to the 4 classes of antiretroviral drugs that meet the defined inclusion and exclusion criteria.

All the clinical centres of Infectious Diseases of the different Italian regions can participate in the implementation of the Registry. Based on an analysis conducted on data collected in an AIFA register, established for the purpose of monitoring the use of dolutegravir (DTG) 50 mg Bis in Die (BID) and containing about 200 patients with the criteria specified in this protocol, the size currently conceivable for this register in Italy is about 300 patients.

The collection of clinical information and biological samples will begin once the Ethics Committee of the participating centers has approved the participation in the registry and will continue for at least three years.

ELIGIBILITY:
Inclusion Criteria:

* subjects with HIV-1 infection;
* age >14 years;
* documented resistance to the 4 classes of antiretroviral drugs (NRTI, NNRTI, PI, INI), defined as resistance (at least intermediate) to at least one of the drugs in each class according to the Stanford algorithm. Resistance can be documented either at the time of inclusion in the study or previously documented throughout the patient's therapeutic history.

Exclusion Criteria:

* none

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Italian PRESTIGIO register will include patients who are regularly monitored according to the principles of good clinical practice in the Italian Infectious Diseases Centres of all Italian regions.
  Patients will be included in the registry once informed consent has been obtained (Annex 2) signed to allow for the recording and analysis of clinical/laboratory data and for the collection of biological samples, subject to the guarantee of anonymity and independence of therapeutic choices and clinical management, which will be the sole responsibility of the treating physician. The consent collected must be entered in the Register.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of date to evaluate: - Long-term effectiveness of different ART; -comorbidity and mortality; - ART compliance and health assessments; - drug-economy indications related to the clinical management. | each 1 year
  to evaluate the characteristics of the study population, will be carry out specific observational studies with the following collected data:
  * demographic characteristics
  * clinical characteristics (HIV transmission mode, pre-ART viral load, CD4+ nadir, co-infection with hepatitis B and C viruses and previous treatments, previous AIDS events);
  * lifestyle factors
  * comorbidity (cancer, diabetes, cardiovascular disease, chronic kidney disease, liver disease, fractures and osteoporosis, cognitive dysfunction, COPD, sexually transmitted diseases);
  * antiretroviral and concomitant drugs;
  * adherence to antiretroviral therapy;
  * Laboratory parameters: CD4, CD8, HIV-RNA, lipids, glucose, liver and kidney parameters;
  * resistance tests for INSTI, NRTI, NNRTI, PI;
  * the historical genotypes (resistance and viral tropism)
  * any hospitalizations;
  * death.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Castagna, Principal Investigator — san raffaele
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in scientific conferences and meetings.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available after 1 year from the first visit first patient (FVFP) and they will be available until patients registry will be updated.
Access Criteria: Must to be a partecipant of the registry.
URL: https://registroprestigio.org/

REFERENCES:
- [Derived] Benlarbi M, Richard J, Clemente T, Bourassa C, Tolbert WD, Prakash M, Chandravanshi M, Clark A, Pazgier M, Durand M, Castagna A, Finzi A. Fostemsavir Decreases the Levels of Anti-gp120 CD4-Induced Antibodies in Heavily Treatment-Experienced People With HIV. J Infect Dis. 2025 Sep 24:jiaf461. doi: 10.1093/infdis/jiaf461. Online ahead of print. PMID 40990223
- [Derived] Clemente T, Galli L, Lolatto R, Gagliardini R, Lagi F, Ferrara M, Cattelan AM, Foca E, Di Biagio A, Cervo A, Calza L, Maggiolo F, Marchetti G, Cenderello G, Rusconi S, Zazzi M, Santoro MM, Spagnuolo V, Castagna A; PRESTIGIO Study Group. Cohort profile: PRESTIGIO, an Italian prospective registry-based cohort of people with HIV-1 resistant to reverse transcriptase, protease and integrase inhibitors. BMJ Open. 2024 Feb 10;14(2):e080606. doi: 10.1136/bmjopen-2023-080606. PMID 38341206
- [Derived] Rusconi S, Saladini F, Bellocchi MC, Galli L, Gagliardini R, Gazzola L, Francisci D, Vichi F, Foca E, Zazzi M, Santoro MM, Gabrieli A, Castagna A; PRESTIGIO Registry study group; PRESTIGIO Registry Steering Committee: Antonella Castagna (coordinator); Stefano Bonora; Leonardo Calza; Antonella Castagna; Giovanni Cenderello; Adriana Cervo; Giulio Maria Corbelli; Antonio Di Biagio; Emanuele Foca; Roberta Gagliardini; Laura Galli; Riccardo Lolatto; Franco Maggiolo; Giulia Marchetti; Stefano Rusconi; Maria Santoro; Vincenzo Spagnuolo; Katia Sterrantino; Maurizio Zazzi. Leronlimab (PRO 140) in vitro activity against 4-class drug resistant HIV-1 from heavily treatment experienced subjects. Pharmacol Res. 2022 Feb;176:106064. doi: 10.1016/j.phrs.2022.106064. Epub 2022 Jan 6. No abstract available. PMID 34999223
- See also: REGISTER E-CRF WEBSITE — https://trials-ice2.advicepharma.com/PRESTIGIO/